CLINICAL TRIAL: NCT06747260
Title: Feasibility and Safety of Intranasal Breast Milk in Hypoxic-ischaemic Encephalopathy
Brief Title: Feasibility and Safety of Intranasally Administered Breast Milk in HIE
Acronym: F-NEO-BRIGHT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SE-NEONAT-03/2024
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Hypoxic Ischaemic Encephalopathy (HIE); Hypoxic Ischemic Encephalopathy of Newborn; Neonatal Encephalopathy; Neonatal Hypoxic Ischemic Encephalopathy; Brain Injury; Perinatal Asphyxia; Perinatal Asphyxia , Moderate to Severe HIE
Keywords: Hypoxic-ischaemic encephalopathy; Neonatal encephalopathy; Perinatal asphyxia; Breast milk; Breast milk stem cells; Intranasal breast milk
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal breast milk (Experimental): Study participants receive their own mother's fresh breast milk, expressed within 4 hours, administered 2 times daily, 0.4 ml in each nostril for 28 days.
  Interventions: Biological: Intranasal breast milk

INTERVENTIONS:
Biological: Intranasal breast milk — Neonates with hypoxic-ischemic encephalopathy receive their own-mother's fresh breast milk intranasally, starting from the first 48 hours of life and continuing for 28 days. Dose: 2 times daily, 0.4 ml in each nostril (15 minutes apart).

SUMMARY:
This is a prospective intervention single center study to evaluate the feasibility and safety of intranasal breast milk in hypoxic-ischaemic encephalopathic neonates receiving therapeutic hypothermia.

DETAILED DESCRIPTION:
Perinatal asphyxia and the resulting hypoxic-ischemic encephalopathy (HIE) are the leading cause of neonatal mortality and long-term neurodevelopmental disabilities. Based on our current knowledge, therapeutic hypothermia is the only therapy that has been proven to reduce central nervous system damage in HIE neonates. Improving neurodevelopmental outcomes of newborns with HIE has been an intense area of research over the past decade.

Breast milk is a complex biological substance that contains a variety of bioactive components including neurotrophic growth factors, cytokines, immunoglobulins, and multipotent stem cells. Studies have shown that exclusive breastfeeding in the early stages of development has a positive impact on cognitive outcomes. Animal studies support that mesenchymal stem cells and neurotrophic substances found in breast milk, when administered intranasally enter the central nervous system and reduce the extent of neurological damage. In preterm infants, it has been shown that intranasally administered breast milk is safe and well-tolerated.

In this prospective study our aim is to assess the feasibility and safety of intranasally delivered breast milk to HIE infants treated with hypothermia. Our objective is to administer fresh, own-mother's breast milk intranasally to neonates with HIE starting from the first day of life and continuing for 1 month.

Feasibility will be based on the ability to initiate treatment within 48 hours of birth using own mother's fresh milk expressed within 4 hours and continuing treatment after discharge until day 28. Safety will be assessed through monitoring vital signs and documenting any adverse events. Time to reach full enteral feeding and lengths of exclusive breast feeding will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe hypoxic- ischaemic encephalopathy, receiving therapeutic hypothermia
* ≥ 35. gestational week
* < 48 hours of life
* Hypothermia treatment for 72 hours
* Parental consent form

Exclusion Criteria:

* Congenital malformation
* Concurrent cerebral lesions
* ECMO therapy
* Contraindication of lactation
* Mother unable or unwilling to provide fresh breast milk
* Postpartum asphyxia

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients where treatment was initiated within 48 hours | 1 months
  Feasibility will be based on the ability to initiate treatment within 48 hours of birth using own mother's fresh milk.

SECONDARY OUTCOMES:
Number of adverse events associated with breast milk administration | 1 month
  Number of adverse events associated with breast milk administration will be recorded, including desaturation (SpO2<80%), bradycardia (heart rate <70% of baseline), apneic episode requiring bag and mask ventilation within 5 minutes of the intervention, or an increase in respiratory support (mode, setting, or FiO2 increase >10%) within 1 hour of the intervention.
Time to reach full enteral feeding | 1 month
  Time to reach full enteral feeding will be recorded and analyzed as a secondary outcome.
Length of exclusive breast feeding | 2 years
  Lengths of exclusive breast feeding will be recorded and analyzed as a secondary outcome.
Total number of treatments during first months of life | 1 months
  Total number of treatments administered in hospital and at home during the first months of life

CONTACTS AND LOCATIONS:
Overall Officials: Unoke Meder, MD, PhD, Principal Investigator — Department of Neonatology, Pediatric Center, Semmelweis University, Budapest, Hungary
Locations (1):
- Division of Neonatology, Pediatric Center, Semmelweis University, Budapest, Hungary, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
On special request pending data transfer agreement approval by Semmelweis University.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 20.12.2024.-01.01.2026.
Access Criteria: Sharing upon reasonable request.
URL: https://semmelweis.hu/bokayklinika/kutatas/asphyxia-munkacsoport/

REFERENCES:
- [Background] Baak LM, Wagenaar N, van der Aa NE, Groenendaal F, Dudink J, Tataranno ML, Mahamuud U, Verhage CH, Eijsermans RMJC, Smit LS, Jellema RK, de Haan TR, Ter Horst HJ, de Boode WP, Steggerda SJ, Prins HJ, de Haar CG, de Vries LS, van Bel F, Heijnen CJ, Nijboer CH, Benders MJNL. Feasibility and safety of intranasally administered mesenchymal stromal cells after perinatal arterial ischaemic stroke in the Netherlands (PASSIoN): a first-in-human, open-label intervention study. Lancet Neurol. 2022 Jun;21(6):528-536. doi: 10.1016/S1474-4422(22)00117-X. PMID 35568047
- [Background] Hoban R, Gallipoli A, Signorile M, Mander P, Gauthier-Fisher A, Librach C, Wilson D, Unger S. Feasibility of intranasal human milk as stem cell therapy in preterm infants with intraventricular hemorrhage. J Perinatol. 2024 Nov;44(11):1652-1657. doi: 10.1038/s41372-024-01982-8. Epub 2024 Apr 30. PMID 38688998
- [Background] Keller T, Korber F, Oberthuer A, Schafmeyer L, Mehler K, Kuhr K, Kribs A. Intranasal breast milk for premature infants with severe intraventricular hemorrhage-an observation. Eur J Pediatr. 2019 Feb;178(2):199-206. doi: 10.1007/s00431-018-3279-7. Epub 2018 Nov 1. PMID 30386923